CLINICAL TRIAL: NCT00319722
Title: Electrophysiologic Indicators of Gating and Timing Abnormalities in Autism
Brief Title: EEG Studies of Sensory Processing in Autistic Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: CURE Foundation (Other); The Commonwealth Fund (Other); National Alliance for Autism Research (Other); Nancy Lurie Marks Family Foundation (Other)
Responsible Party: Katherine M. Martien, M.D., Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2005-P-000868/3
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-05

CONDITIONS: Autism
Keywords: autism; pervasive developmental disorder; evoked potentials; EEG; Coherence
MeSH Terms: conditions — Autistic Disorder; Child Development Disorders, Pervasive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
This study uses EEG to study brain waves at rest and in response to specific auditory and visual sensory stimuli in autistic children. We hypothesize that, compared to same age peers, autistics will show abnormalities in their electrophysiologic processing of sounds (tones and phonemes)and visual stimuli (flashes of light)and that these abnormalities will be able to separate autistics not only from typical children but also into clinical subgroups with specific biological/electrophysiological characteristics. We hope to find biological measures which will prove diagnostic of autism in very young children and which can be used in the measurement of treatment outcome in future intervention trials.

DETAILED DESCRIPTION:
Specific Aims:

Aim 1: To recruit 75 children with autism and 75 age- and sex-matched controls ages 6 to 8 years old for an electrophysiological study and to characterize the subjects using appropriate instruments for autism diagnosis, language functioning and behavior/sensory profile, and to measure head circumferences Aim 2: To acquire and analyze event-related potential (ERP) data in the auditory and visual modality.

ERP Hypothesis: Increased amplitude, altered morphology, impaired temporal discrimination and delayed responsiveness will be found early in the processing hierarchy, and the severity of these abnormalities will be associated with the severity of dysfunction at higher levels of cortical processing.

Aim 3: To acquire EEG data and to analyze it quantitatively. Quantitative EEG Hypothesis: Both interhemispheric and intrahemispheric coherence measures of the EEG will be significantly deviant from those in the normal sample and predicted by abnormalities of ERPs. In addition, EEG background alpha activity will show post mature (i.e. higher) frequencies (Hz) than would be expected for age and focal epileptiform activity and slowing (i.e. paroxysmal theta) will predict dysfunction on the ERPs.

Rationale:

The goal of this grant is to use electrophysiological measures to characterize abnormalities in gating and timing in the autistic brain. The motivation for this research project derives from findings and models in autism of increased excitation/inhibition ratios, increased brain and white matter volume and altered connectivity. These changes, alone and in combination, have the potential to alter the intensity, timing and integration of signaling at multiple stages of processing. These signaling problems can potentially lead to the autistic behavioral phenotype through cognitive processing abnormalities including the hyperspecificity/overselectivity of autism, as well as to such features of autism as sensory processing abnormalities, seizures, and anxiety. We believe that characterizing abnormalities related to gating and timing phenomena may lead to the development of an electrophysiological battery that can be utilized for early diagnosis, prognosis and subtyping of autism, as well as the tracking of treatment efficacy.

Subjects:

Subjects will be recruited from the general population, the Ladders Clinic at MGH/Spaulding Hospital, where the PI, Dr. Martien, is employed as a clinician, as well as from the clinical practice of Dr. Herbert at the MGH-Institute of Health Professions preschool clinic. Flyers will be placed on available bulletin boards at the two clinics and throughout the greater Boston area, particularly at all Partners, Harvard, MIT, hospital, clinic, research, and educational settings.

The study will seek to enroll eighty 75, 6 to 8 year olds with autism and 75 age and sex matched controls. Children will be considered for inclusion in the autism group if:

* English is the primary language in the home
* Experimental group: Child meets criteria for autism on the ADI-R and ADOS evaluation scales (this inclusion criteria will be explained during the consent process).

They meet non of the Exclusionary criteria, which include:

* Known genetic disorder
* Hearing or gross sensorimotor deficits
* Clinical evidence of progressive encephalopathy
* Asphyxia at birth or any other time
* Frequent seizures or use of anticonvulsant drugs or psychotropic medication
* Known presence of focal brain lesions, brain atrophy or ventriculomegaly. Children will be considered for the control group if the child meets all of the above criteria except they do not meet the criteria for autism or close to it on the ADOS and ADI-R evaluation scales.

Methods:

The child will be seated in a comfortable chair and the physiological assessment will begin after a head circumference is obtained with a tape measure, an EEG cap is placed on the child's head and gel is applied to each electrode in the cap. The tasks include 5 minutes of baseline EEG recording while the child is looking at a design on a monitor placed 2 meters in front of the chair. We then will proceed with a series of auditory and visual stimuli presented by computer through two speakers placed 1 meter in front of the child (auditory) and strobe (visual) at 50 cm. The paradigms will include a presentation of pairs of tones with variable interstimulus intervals presented in random order at 65 dB SPL, a paradigm with either 1000 Hz or 800 Hz at 65 dB, and a final auditory paradigm with two different phonemes, presented at 65 dB. The visual tasks will involve the presentation of flashes of light which vary in frequency and luminance both reflected off a white board one meter from the child and directly at the child's visual field. In each series, there will be a 1 minute break between two blocks of 100 trials each for a total of 200 trials. The experimenter will show the child an interesting toy and talk to the child during the break.

The parent will be asked to complete the Vineland Adaptive Behavior Scales, the Communication and Symbolic Behavior Scales (CSBS) and the MacArthur Communicative Development Inventory. In the case that the subjects are recruited from the Ladders infant sib study, we will use the existing ADI-R and ADOS data because Ladders has authorized the release of this information.

The total time for the laboratory session will be approximately 1 hour. The full battery of tasks will be performed on compliant children. For those children whose attention cannot be maintained for the full battery, the examiner will stop and give breaks as needed. The examiner will go on to the next task or terminate the session if the subject or parent of the subject chooses to do so.

ELIGIBILITY:
Inclusion Criteria:

autistic children or their younger siblings between the ages of 3 months to 8 year

Controls: typically developing children 3mo to 8 years without known language or social disorder and not related to child with autism

Exclusion Criteria: progressive encephalopathy, treatment with multiple antiepileptic drugs, known genetic diagnosis.

-

Ages: 3 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: autistic children meeting criteria for autism based on ADOS and ADI and clinical DSM IV or their siblings between the ages of 3 months to 13 years.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2006-02; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
EEG and ERP abnormalities | 2 years

SECONDARY OUTCOMES:
Characteristic and severity of autistic behaviors | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M. Martien, M.D., Principal Investigator — Massachusetts General Hospital; Martha Herbert, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH LADDERS Clinic, Lexington, Massachusetts, United States